CLINICAL TRIAL: NCT04133064
Title: Pivot Breath Sensor Study to Evaluate the Effect of the Pivot Breath Sensor on a User's Attitudes Towards Quitting Smoking and Smoking Behavior.
Brief Title: Assessment of the Pivot Breath Sensor: Single-Arm Cohort Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jennifer Marler, MD (Industry)
Responsible Party: Sponsor-Investigator, Jennifer Marler, MD, Senior Director, Clinical and Medical Affairs, Pivot Health Technologies Inc.
Organization: Pivot Health Technologies Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: c-202
Record Dates: First submitted 2019-10-09; First posted 2019-10-21 (Actual); Results first posted 2022-11-09 (Actual); Last update posted 2022-11-09 (Actual); Status verified 2022-10

CONDITIONS: Smoking Reduction; Smoking Behaviors; Smoking, Tobacco; Smoking Cessation
MeSH Terms: conditions — Smoking Reduction; Smoking; Tobacco Smoking; Smoking Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Pivot Breath Sensor (user group) (Other): Self-reported daily smokers of 10 or more cigarettes per day
  Interventions: Device: Pivot Breath Sensor

INTERVENTIONS:
Device: Pivot Breath Sensor — The Pivot Breath Sensor measures the level of carbon monoxide in exhaled breath and displays the carbon monoxide value to the user.

SUMMARY:
Prospective open label, single center study enrolling up to 220 participants to evaluate the effect of the Pivot Breath Sensor on a user's attitudes towards quitting smoking and smoking behavior.

DETAILED DESCRIPTION:
Study to collect the following data during and after use of a personal carbon monoxide breath sensor (Pivot Breath Sensor):

* Change in attitudes towards quitting smoking
* Change in smoking behavior
* Participant feedback

ELIGIBILITY:
Inclusion Criteria:

* 18-80 years of age
* Current daily cigarette smokers (at least 10 cigarettes per day)
* Resident of the United States
* Able to read and comprehend English
* Owns and uses a smartphone compatible with the study app (iPhone 5 and above with operating system iOS 11 and above, or, Android 5.0 and above with operating system Android 5.0 and above)
* Willing to sign the Informed Consent Form

Exclusion Criteria:

* Pregnancy
* Participation in a previous study sponsored by Carrot Inc

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 234 (Actual)
Dates: Start 2019-09-25 (Actual); Primary Completion 2020-03-10 (Actual); Study Completion 2020-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jen Marler, Principal Investigator — Pivot Health Technologies Inc.
Locations (1):
- Carrot Inc., Redwood City, California, United States

REFERENCES:
- [Derived] Marler JD, Fujii CA, Wong KS, Galanko JA, Balbierz DJ, Utley DS. Assessment of a Personal Interactive Carbon Monoxide Breath Sensor in People Who Smoke Cigarettes: Single-Arm Cohort Study. J Med Internet Res. 2020 Oct 2;22(10):e22811. doi: 10.2196/22811. PMID 32894829

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Pivot Breath Sensor (User Group)
Started | 234
Completed | 215
Not Completed | 19

BASELINE CHARACTERISTICS:
Population: Participants that enrolled in the study and completed the baseline questionnaire.
Arm/Group | Pivot Breath Sensor (User Group)
Number analyzed (Participants) | 234
Age, Customized [Count of Participants; unit: Participants]
  18-29 years | 37
  30-60 years | 185
  61-80 years | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123
  Male | 111
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White | 209
  Race/Ethnicity: Hispanic, Latinx, or Spanish Origin | 5
  Race/Ethnicity: Black or African American | 9
  Race/Ethnicity: Asian | 3
  Race/Ethnicity: American Indian or Alaska Native | 2
  Race/Ethnicity: Middle Eastern or North African | 1
  Race/Ethnicity: Hawaiian or Other Pacific Islander | 0
  Race/Ethnicity: Some other race, ethnicity, or origin | 5
  Race/Ethnicity: Prefer not to answer | 0
Region of Enrollment [Number; unit: participants]
  United States | 234
Education [Count of Participants; unit: Participants]
  Less than 8th grade | 0
  Some high school | 7
  High school/General educational development | 50
  Some college | 107
  Associate's (2-year) degree | 37
  Bachelor's (4-year) degree | 25
  Master's degree | 7
  Professional or doctorate degree | 1
Employment [Count of Participants; unit: Participants]
  Unemployed | 11
  Employed <20 hours/week | 29
  Employed ≥ 20 hours/week | 194
Years smoking [Mean (Standard Deviation); unit: years] | 21.7 (11.5)
Cigarettes per day (CPD) [Mean (Standard Deviation); unit: cigarettes smoked per day] | 20.3 (8)
Would you like to stop smoking? [Count of Participants; unit: Participants]
  yes | 217
  no | 17
Motivation to Quit (Stage of Change) - Are you seriously thinking of quitting smoking? [Count of Participants; unit: Participants]
  Yes, within the next 30 days | 36
  Yes, within the next 6 months | 180
  No, not thinking of quitting | 18
Readiness to Quit (RTQ) [Mean (Standard Deviation); unit: units on a scale] — How ready are you to quit smoking? Answered on a 1-10 scale: 1 = Not at all ready; 10 = Completely ready
  units on a scale | 5.6 (2.7)
Success to quit (STQ) [Mean (Standard Deviation); unit: units on a scale] — If you were to quit smoking right now, how successful would you be? Answered on a scale: 1 = Not at all successful; 10 = Completely successful
  units on a scale | 3.3 (2.3)
Difficulty to quit (DTQ) [Mean (Standard Deviation); unit: units on a scale] — If you were to quit smoking right now, how difficult do you think it would be to stay smoke free? Answered on a scale: 1 = Really hard to stay quit; 10 = Really easy to stay quit
  units on a scale | 2.8 (2.4)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Different Stages of Change in Desire to Quit Smoking
Description: Assessment of participant's desire to quit by measuring Stage of Change.
  The participant will be asked if they are serious about quitting smoking and they can select from the following options:
  * Yes, within the next 30 days
  * Yes, within the next 6 months
  * No, not thinking of quitting All data obtained via questionnaires completed by the participants. Throughout the course of the study, if the participant moves from "No, not thinking of quitting" to "yes, within the next 6 months" to "Yes, within the next 30 days" - that is a positive outcome for the participant. If they answered in the reverse, that would be a negative outcome for the participant. In short, becoming more ready to quit is a positive outcome, becoming less ready to quit is a less positive outcome.
Time Frame: 3 months (12 weeks) compared to baseline
Population: Participants that completed the 12-week questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Pivot Breath Sensor (User Group)
Number analyzed (Participants) | 215
Participants
  Increased motivation to quit | 84
  Unchanged motivation to quit | 118
  Decreased motivation to quit | 13

2. Primary Outcome: Success to Quit (STQ)
Description: Assessment of participant's attitudes towards quitting by measuring Success to Quit.
  The participant will be asked If you were to quit smoking right now, how successful would you be? Rating Scale: 1 = Not at all successful, 10 = Completely successful. Higher score is a better outcome for participants, it indicates a more positive attitude towards quitting smoking.
Time Frame: 3 months (12 weeks)
Population: Participants that completed the 12 week questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pivot Breath Sensor (User Group)
Number analyzed (Participants) | 215
units on a scale | 5 (3.1)

3. Primary Outcome: Difficulty to Quit (DTQ)
Description: Assessment of participant's attitudes towards quitting by measuring Perceived Difficulty to staying Quit.
  Participant will be asked: If you were to quit smoking right now, how difficult do you think it would be to stay smoke free? Rating scale: 1 = Really hard to stay quit, 10 = Really easy to stay quit. Higher score is a better outcome for participants, it indicates a more positive attitude towards quitting smoking, specifically lower perceived difficulty to quit.
Time Frame: 3 months (12 weeks)
Population: Participants that completed the 12 week questionnaire
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Pivot Breath Sensor (User Group)
Number analyzed (Participants) | 215
units on a scale | 4.3 (3.0)

4. Primary Outcome: Average Quit Attempts Made Since Using the Pivot Breath Sensor
Description: Assess participant's smoking behavior by measuring Quit attempts. Participant were asked: Since you began using the Pivot Breath Sensor, how many times have you tried to quit smoking?
Time Frame: 3 months (12 weeks)
Population: Participants that completed the 12 week questionnaire
Measure: Mean (Standard Deviation); unit: quit attempts made
Arm/Group | Pivot Breath Sensor (User Group)
Number analyzed (Participants) | 215
quit attempts made | 2.4 (9.1)

5. Primary Outcome: Change in Cigarettes Per Day (CPD) From Baseline
Description: Assess participant's smoking behavior by measuring CPD. Participant will be asked to enter a number for: How many cigarettes do you now smoke per day, on average? Enter number value.
Time Frame: 3 months (12 weeks)
Population: Participants that completed the 12 week questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Pivot Breath Sensor (User Group)
Number analyzed (Participants) | 215
Participants
  Reduced CPD from baseline | 178
  No change in CPD from baseline | 25
  Increased CPD from baseline | 12

6. Primary Outcome: Point Prevalence Abstinence (PPA)
Description: Assess participant's smoking behavior by measuring 7-Day and 30-Day PPA. Participant will be asked: In the last 7 days and 30 days have you smoked any cigarettes? Answer choice: Yes/No 7-Day PPA is defined as answering "No" to "In the last 7 days have you smoked any cigarettes?" 30-Day PPA is defined as answering "No" to "In the last 30 days have you smoked any cigarettes?" Data obtained via questionnaires completed by the participants.
Time Frame: 3 months (12 weeks)
Population: Participants that completed the 12 week questionnaire
Measure: Count of Participants; unit: Participants
Groups:
- Pivot Breath Sensor (User Group) - Intention to Treat (ITT): Participants that enrolled and completed the baseline questionnaire
  Self-reported daily smokers of 10 or more cigarettes per day
  Pivot Breath Sensor: The Pivot Breath Sensor measures the level of carbon monoxide in exhaled breath and displays the carbon monoxide value to the user.
- Pivot Breath Sensor (User Group) - Completer: Participants that completed the 12 week questionnaire
  Self-reported daily smokers of 10 or more cigarettes per day
  Pivot Breath Sensor: The Pivot Breath Sensor measures the level of carbon monoxide in exhaled breath and displays the carbon monoxide value to the user.
Arm/Group | Pivot Breath Sensor (User Group) - Intention to Treat (ITT) | Pivot Breath Sensor (User Group) - Completer
Number analyzed (Participants) | 234 | 215
Participants
  7-day PPA | 28 | 28
  30-day PPA | 14 | 14

7. Secondary Outcome: Feedback on Breath Sensor Setup, Experience and Use
Description: Gather participant feedback on breath sensor setup:
  Participant is asked:
  1. How would you rate the ease or difficulty of getting started with the breath sensor?
  2. How would you rate the ease or difficulty of following the directions on the breath sensor screen?
  3. If you ever got an error on the breath sensor screen, how easy or difficult was it to understand the issue and correct it?
  Select one:
  1. - Very difficult
  2. - Difficult
  3. - Neither easy nor difficult
  4. - Easy
  5. - Very Easy I did not set up my breath sensor All data obtained via questionnaires completed by the participants.
Time Frame: 1 week
Population: Participants that completed the 1 week questionnaire. For question 3: If you ever got an error on the breath sensor screen, how easy or difficult was it to understand the issue and correct it? Other category = "I set up my breath sensor but have not gotten an error on the breath sensor screen"
Measure: Count of Participants; unit: Participants
Arm/Group | Pivot Breath Sensor (User Group)
Number analyzed (Participants) | 227
Participants
  How would you rate the ease or difficulty of getting started with the breath sensor?: 1 - Very Difficult | 1
  How would you rate the ease or difficulty of getting started with the breath sensor?: 2 - Difficult | 9
  How would you rate the ease or difficulty of getting started with the breath sensor?: 3 - Neither easy nor difficult | 10
  How would you rate the ease or difficulty of getting started with the breath sensor?: 4 - Easy | 42
  How would you rate the ease or difficulty of getting started with the breath sensor?: 5 - Very easy | 165
  How would you rate the ease or difficulty of getting started with the breath sensor?: Other | 0
  How would you rate the ease or difficulty of following the directions on the breath sensor screen?: 1 - Very Difficult | 1
  How would you rate the ease or difficulty of following the directions on the breath sensor screen?: 2 - Difficult | 0
  How would you rate the ease or difficulty of following the directions on the breath sensor screen?: 3 - Neither easy nor difficult | 7
  How would you rate the ease or difficulty of following the directions on the breath sensor screen?: 4 - Easy | 36
  How would you rate the ease or difficulty of following the directions on the breath sensor screen?: 5 - Very easy | 183
  How would you rate the ease or difficulty of following the directions on the breath sensor screen?: Other | 0
  If you ever got an error ... how easy or difficult was it to understand the issue and correct it?: 1 - Very Difficult | 0
  If you ever got an error ... how easy or difficult was it to understand the issue and correct it?: 2 - Difficult | 5
  If you ever got an error ... how easy or difficult was it to understand the issue and correct it?: 3 - Neither easy nor difficult | 8
  If you ever got an error ... how easy or difficult was it to understand the issue and correct it?: 4 - Easy | 37
  If you ever got an error ... how easy or difficult was it to understand the issue and correct it?: 5 - Very easy | 92
  If you ever got an error ... how easy or difficult was it to understand the issue and correct it?: Other | 85

8. Secondary Outcome: Feedback on Impact on Motivation to Quit Smoking
Description: Gather participant feedback on impact of breath sensor:
  Participant will be asked: How has using the breath sensor affected your motivation to quit smoking?
  Select one:
  * Using the breath sensor has increased my motivation to quit smoking
  * Using the breath sensor has not affected my motivation to quit smoking
  * Using the breath sensor has decreased my motivation to quit smoking
  * I haven't used the breath sensor
Time Frame: 1 week
Population: Participants that completed the 1 week questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Pivot Breath Sensor (User Group)
Number analyzed (Participants) | 227
Participants
  Using the breath sensor has increased my motivation to quit smoking | 171
  Using the breath sensor has not affected my motivation to quit smoking | 55
  Using the breath sensor has decreased my motivation to quit smoking | 0
  I haven't used the breath sensor | 1

9. Secondary Outcome: Feedback on Impact on Number of Cigarettes Smoked Per Day
Description: Gather participant feedback on impact of breath sensor:
  Participant will be asked: How has using the breath sensor affected the number of cigarettes you smoke per day?
  Select one:
  * Using the breath sensor has increased the number of cigarettes I smoke per day
  * Using the breath sensor has not affected the number of cigarettes I smoke per day
  * Using the breath sensor has decreased the number of cigarettes I smoke per day
  * I haven't used the breath sensor
Time Frame: 1 week
Population: Participants that completed the 1 week questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Pivot Breath Sensor (User Group)
Number analyzed (Participants) | 227
Participants
  Using the breath sensor has increased the number of cigarettes I smoke per day | 2
  Using the breath sensor has not affected the number of cigarettes I smoke per day | 119
  Using the breath sensor has decreased the number of cigarettes I smoke per day | 105
  I haven't used the breath sensor | 1

10. Secondary Outcome: Feedback on Commercialization
Description: Gather participant feedback on commercialization:
  Participant will be asked: Hypothetical: if it was commercially available, would you be interested in buying the Pivot Breath Sensor? Answer: Yes/No
Time Frame: 4 weeks
Population: Participants that completed the 4 week questionnaire
Measure: Count of Participants; unit: Participants
Arm/Group | Pivot Breath Sensor (User Group)
Number analyzed (Participants) | 216
Participants
  yes | 153
  no | 63

ADVERSE EVENTS:
Time Frame: Adverse events were assessed for over 12 weeks
Arm/Group | Pivot Breath Sensor (User Group)
All-Cause Mortality (participants affected / at risk) | 0/234
Serious Adverse Events (participants affected / at risk) | 0/234
Other Adverse Events (participants affected / at risk) | 0/234

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-09-12): https://cdn.clinicaltrials.gov/large-docs/64/NCT04133064/Prot_SAP_001.pdf